CLINICAL TRIAL: NCT06554288
Title: Pharmacogenomic Contribution to the Biotransformation of Trihexyphenidyl and Development of a Precision Dosing Model for Children With Dystonia and Cerebral Palsy
Brief Title: Pharmacogenomic Contributions to Trihexyphenidyl Biotransformation and Response in Children With Dystonic Cerebral Palsy
Acronym: TRIKE2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Rose Gelineau-Morel, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003228
Record Dates: First submitted 2024-07-29; First posted 2024-08-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Disorder; Genetic Predisposition; Dystonia, Secondary; Dystonia; Cerebral Palsy, Dystonic-Rigid; Cerebral Palsy, Dyskinetic; Trihexyphenidyl Adverse Reaction; Pharmacogenomic Drug Interaction
Keywords: Pediatric; Cerebral Palsy; Dystonia; Pharmacogenomics; Trihexyphenidyl
MeSH Terms: conditions — Genetic Predisposition to Disease; Dystonic Disorders; Dystonia; Cerebral Palsy | interventions — Trihexyphenidyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trihexyphenidyl (Experimental): Participants receive trihexyphenidyl following the dose escalation schedule below:
  Week 1: 0.05 mg/kg BID Week 2: 0.05 mg/kg TID Week 3: 0.1 mg/kg TID Week 4: 0.15 mg/kg TID Week 5: 0.20 mg/kg TID Week 6-15: 0.25 mg/kg TID
  Interventions: Drug: Trihexyphenidyl

INTERVENTIONS:
Drug: Trihexyphenidyl — 6-week dose escalation up to 0.25mg/kg TID, followed by a 9-week maintenance period at this dose

SUMMARY:
This study looks at how a medicine called trihexyphenidyl works in children with dystonic cerebral palsy. The study aims to understand how trihexyphenidyl is broken down and used in the body of pediatric patients and whether this is impacted by a person's genetics. Information from this study will also be used to design future clinical trials.

DETAILED DESCRIPTION:
This is a 16-week single-arm nonrandomized pilot study of trihexyphenidyl in children with dystonic cerebral palsy (DCP) to 1) evaluate the pharmacokinetics (PK) of trihexyphenidyl (THP) and variation in PK parameters between CYP2D6 and CYP2C19 genotypes and 2) evaluate the feasibility of a future exposure-controlled clinical trial of THP.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5-17 years of age
* Diagnosis of cerebral palsy and dystonia causing interference
* Parent/legal guardian of a child with a diagnosis of cerebral palsy and dystonia
* Parent/legal guardian is willing and able to provide informed permission/assent for the study

Exclusion Criteria:

* Previously or currently taking trihexyphenidyl
* Patients turning 18 years of age within the study period (16 weeks from Study Day 1)
* A language barrier for the patient that precludes communication and/or the ability to complete study-related requirements

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Cmax between CYP2D6 and CYP2C19 phenotype groups | Baseline
  Cmax will be measured in first-dose pharmacokinetic study on study day 1
Difference in AUC0-n between CYP2D6 and CYP2C19 phenotype groups | Baseline
  AUC0-n will be measured in first-dose pharmacokinetic study on study day 1
Difference in AUC0-∞ between CYP2D6 and CYP2C19 phenotype groups | Baseline
  AUC0-∞ will be measured in first-dose pharmacokinetic study on study day 1
Recruitment percentage | Through study completion, an average of 2 years
  Measure percent of participants who were approached for the study that enrolled in the study
Retention percentage | Through study completion, an average of 2 years
  Measure percent of participants enrolled who completed the study
Dystonia Efficacy Measures Outcome Completion | Through study completion, an average of 2 years
  Measure percent of participants enrolled who were able to complete each dystonia efficacy measure (see secondary outcome measures)

SECONDARY OUTCOMES:
Number of participants with at least one adverse event as measured by the Safety Monitoring Uniform Report Form (SMURF) | Through study completion, an average of 2 years
  Adverse events will only include those that are determined to be related to the study drug.
Change from baseline in dystonia duration as measured by the Dyskinesia Impairment Scale (exploratory) | Baseline, 16 weeks
  Duration of dystonia using subscale DIS-D are measured in 12 body regions during activity and rest.
  Dystonia duration scores are measured on a 4-point scale from 0 to 4 with 0 being dystonia is absent and 4 being dystonia is always present (≥90%).
Change from baseline in dystonia amplitude as measured by the Dyskinesia Impairment Scale (exploratory) | Baseline, 16 weeks
  Amplitude of dystonia using subscale DIS-D are measured in 12 body regions during activity and rest.
  Dystonia amplitude scores are measured on a 4-point scale from 0 to 4 with 0 being dystonia is absent and 4 being dystonia in maximal range of motion (≥90%).
Change from baseline in dystonia as measured by the Quality of Upper Extremity Skills Test (QUEST) (exploratory) | Baseline, 16 weeks
  Upper extremity function in 1 domain; grasp. 13 activities with item-level scores and three items for the tester to rate: hand function, spasticity, and cooperativeness. All scores are summed, and formulas are used to calculate percentages for this domain. Domain percentage is summed with a minimum score less than 0, and the maximum score is 100.
Change in functional impact from baseline as measured by the Dyskinetic Cerebral Palsy Functional Impact Scale (D-FIS) (exploratory) | Baseline, 16 weeks
  Functional impact scores are measured on a 5-point scale from 0 to 4 with 0 being dyskinesia may be present but has no impact on the named activity, and 4 being dyskinesia is present and prevents child from doing a named activity, even with help. An "NA" option indicates the activity is difficult but NOT due to dyskinesia.
Change in priority scores in functional impact from baseline as measured by the Dyskinetic Cerebral Palsy Functional Impact Scale (D-FIS) (exploratory) | Baseline, 16 weeks
  Priority scores are measured on a 4-point scale from 1 to 4 with 1 being an activity is not a priority and 4 being an activity is highest priority.
Change in patient-driven performance from baseline as measured by the Canadian Occupational Performance Measure (exploratory) | Baseline, 16 weeks
  Performance scores are measured on a 10-point scale with 1 being not able to do an activity at all and 10 being able to do an activity extremely well.
Change in patient-driven goal satisfaction from baseline as measured by the Canadian Occupational Performance Measure (exploratory) | Baseline, 16 weeks
  Satisfaction scores are measured on a 10-point scale with 1 being not satisfied at all with the way they do an activity to 10 being extremely satisfied with the way they do an activity.
Change in caregiver's perspective about their child in 4 domains: health status, comfort, wellbeing, functional abilities, and ease of caregiving from baseline as measured by Caregiver Priorities and Child Health Index of Life with Disabilities | Baseline, 16 weeks
  Scores for each domain and for the total survey are standardized and range from 0 to 100 with 0 being the worst and 100 being the best.
Measure the acceptability of outcome measures at 16 weeks as measured by the Acceptability of Intervention Measure | 16 weeks
  Scores are measured on a 5-point scale from Completely Disagree to Completely Agree for items 1) The outcome measure meets my approval. 2) The outcome measure is appealing to me. 3) I like the outcome measure. 4) I welcome the outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Rose Gelineau-Morel, MD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Hospital Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Pharmacokinetic data, including genotypes and THP levels, will be in publications for analysis replication. This will include participant genotypes and corresponding levels of THP, R-THP, and S-THP. Raw data and technical duplicates are available on request for result transparency and clinical trial design. CYP2D6 and CYP2C19 data will also be published; raw sequences go to NICHD's Data Hub (https://dash.nichd.nih.gov/), new haplotypes to PharmVar (https://www.pharmvar.org/). Recruitment, retention, and scientific methods outcomes will be published to guide future THP trials, though the study isn't powered for efficacy endpoints.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available at the time of the associated publication or at the end of the study period, whichever comes first. The datasets made available through publications in PubMed will be made available indefinitely. Sharing of raw data upon request will be accommodated for at least 10 years. Once genetic data are published or uploaded to DASH or PharmVar, they will be available indefinitely.
Access Criteria: Access to raw pharmacokinetic data/samples and genetic samples will be controlled because it will only be available upon request. For DASH, a request for study data can be submitted and managed within their system.
URL: https://dash.nichd.nih.gov/